CLINICAL TRIAL: NCT04842357
Title: Imparting of Practical Skills by Digital Methods - Effectivity of Digital Education Under Conditions of the Pandemia Concerning the Application of Donati Suture and the Application of an Intraosseous Venous Access
Brief Title: Imparting of Practical Skills by Digital Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Thomas Ott, Thomas Ott, M.D., DESA, Scientific consultant of the simulation center, Department of Anesthesiology, University Hospital Center, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UM-Nr. 21-00483
Record Dates: First submitted 2021-04-06; First posted 2021-04-13 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Clinical Skills; Intra-osseous; Sutures; Education
Keywords: clinical skills; intraosseous access; Donati suture; imparting skills; education; undergraduate education

STUDY DESIGN:
Intervention Model Description: The investigators will recruit last year medical students and randomise them into two groups: Group A and Group B. Both groups will be video recorded during the performance of the two skills on simulators (i.s. Donati suture and intraosseous venous access) (timepoint: T0). Then group A will watch a standardised video about the skills, and group B will do self-study. Then, both groups will be again video recorded during the performance of the two skills on simulators (timepoint: T1). After 1 week group B will watch the same standardised video about the skills, and group A will do self-study. Then both groups will be again video recorded during the performance of the two skills on simulators (timepoint: T2).
Masking Description: The participant cannot be masked because they realise if they are in group A or B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video - then self-study (Other): Group A will be video recorded during the performance of the two skills on simulators (i.e. Donati suture and intraosseous venous access) (timepoint: T0). Then group A will watch a standardised video about the skills, then will be again video recorded during the performance of the two skills on simulators (timepoint: T1). After 1 to 2 weeks group A will do self-study, then will be again video recorded during the performance of the two skills on simulators (timepoint: T2).
  Interventions: Other: standardised video concerning clinical skill
- self-study, then video (Other): Group B will be video recorded during the performance of the two skills on simulators (i.e. Donati suture and intraosseous venous access) (timepoint: T0). Then group B will do self-study, then will be again video recorded during the performance of the two skills on simulators (timepoint: T1). After 1 to 2 weeks group B will watch the standardised video about the skills, then will be again video recorded during the performance of the two skills on simulators (timepoint: T2).
  Interventions: Other: standardised video concerning clinical skill

INTERVENTIONS:
Other: standardised video concerning clinical skill — watching a video concerning clinical skills.

SUMMARY:
Due to the corona pandemia and the consecutive reduction of teaching students face to face the imparting of medical skills is limited. Video sequences may be an adequate alternative to educate selected practical skills. So, the investigators intend to explore this aspect as a first concerning two basic medical skills: Donati suture and intraosseous venous access.

DETAILED DESCRIPTION:
The investigators will recruit last year medical students and randomise them into two groups: Group A and Group B. Both groups will be video recorded during the performance of the two skills on simulators (i.s. Donati suture and intraosseous venous access) (timepoint: T0). Then group A will watch a standardised video about the skills, and group B will do self-study. Then, both groups will be again video recorded during the performance of the two skills on simulators (timepoint: T1). After 1 week group B will watch the same standardised video about the skills, and group A will do self-study. Then both groups will be again video recorded during the performance of the two skills on simulators (timepoint: T2).

ELIGIBILITY:
Inclusion Criteria:

* medical student in the last year of the curriculum

Exclusion Criteria:

* no medical student in the last year of the curriculum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Donati suture: "Task-Specific Score" | 1 week
  Score to quantify the particular skill: Minimum / worst performance 8, Max / best performance: 40
Intraosseous venous access: "Intraosseous Access Performance Assessment Scale" | 1 week
  Score to quantify the particular skill: Minimum / worst performance 0, Max / best performance: 17

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Oliver O. Dietz, M.D., Ph.D., Study Director — Trauma Surgery / Zentrum für Orthopädie und Unfallchirurgie, Langebeckstr. 1, 55131 Mainz, Germany; Thomas Ott, M.D., Study Director — Department of Anaesthesiology / Klinik für Anästhesiologie, Langenbeckstr. 1, 55131 Mainz, Germany
Locations (1):
- University Hospital Centre Mainz, Mainz, RLP, Germany

IPD SHARING:
Plan to Share IPD: Yes
We will decide after ethical review board approval.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: expected 2022
Access Criteria: via journal access policies

REFERENCES:
- [Background] Levitan RM, Bortle CD, Snyder TA, Nitsch DA, Pisaturo JT, Butler KH. Use of a battery-operated needle driver for intraosseous access by novice users: skill acquisition with cadavers. Ann Emerg Med. 2009 Nov;54(5):692-4. doi: 10.1016/j.annemergmed.2009.06.012. Epub 2009 Jul 29. PMID 19643511
- [Background] Lee JC, Boyd R, Stuart P. Randomized controlled trial of an instructional DVD for clinical skills teaching. Emerg Med Australas. 2007 Jun;19(3):241-5. doi: 10.1111/j.1742-6723.2007.00976.x. PMID 17564692
- [Result] Shippey S, Handa VL, Chen TL, Chou B, Bowen CW. Validation of an instrument for evaluation of subcuticular suturing using a plastic tissue model. J Surg Educ. 2009 Jan-Feb;66(1):31-4. doi: 10.1016/j.jsurg.2008.09.001. PMID 19215895
- [Result] Shippey SH, Chen TL, Chou B, Knoepp LR, Bowen CW, Handa VL. Teaching subcuticular suturing to medical students: video versus expert instructor feedback. J Surg Educ. 2011 Sep-Oct;68(5):397-402. doi: 10.1016/j.jsurg.2011.04.006. Epub 2011 Jun 25. PMID 21821220
- [Result] Oriot D, Darrieux E, Boureau-Voultoury A, Ragot S, Scepi M. Validation of a performance assessment scale for simulated intraosseous access. Simul Healthc. 2012 Jun;7(3):171-5. doi: 10.1097/SIH.0b013e31824a5c20. PMID 22511182
- [Derived] Ott T, Demare T, Mohrke J, Silber S, Schwab J, Reuter L, Westhphal R, Schmidtmann I, Dietz SO, Pirlich N, Ziebart A, Engelhard K. Does an instructional video as a stand-alone tool promote the acquisition of practical clinical skills? A randomised simulation research trial of skills acquisition and short-term retention. BMC Med Educ. 2024 Jul 2;24(1):714. doi: 10.1186/s12909-024-05714-6. PMID 38956562